CLINICAL TRIAL: NCT07386860
Title: Randomized Controlled Study on the Effectiveness of Steroid Nasal Drops in the Olfactory Cleft Combined With Olfactory Training for Patients With Post-infectious Olfactory Dysfunction
Brief Title: The Effectiveness of Steroid Nasal Drops in the Olfactory Cleft Combined With Olfactory Training for Patients With PIOD
Acronym: PIOD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dawei Wu, Associate Researcher, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9059106
Record Dates: First submitted 2026-01-24; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Smell Dysfunction
Keywords: post-infectious olfactory dysfunction; olfactory training; steroid drops; combined therapy
MeSH Terms: conditions — Olfaction Disorders | interventions — Olfactory Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hormone Nasal Drops Combined with Olfactory Training Group (Experimental): Olfactory Cleft Steroid Nasal Drops: Patients will be instructed to assume the Mygind position. Five drops of budesonide suspension (2ml:1mg) will be instilled into each nostril to facilitate delivery to the olfactory cleft. This position will be maintained for 5 minutes, after which patients should expectorate any residual medication. The treatment regimen will follow a tapered schedule: twice daily during the first treatment month, reduced to once daily in the second month, and further reduced to every other day in the third month.
  Olfactory Training: Participants will perform olfactory training using a modified training device programmed with four distinct odorants (rose, peppermint, tea tree, and clove). Each odorant will be sniffed for 10 seconds per nostril, with 10-second intervals between odorants. Each training session lasts 5 minutes and is conducted twice daily, before breakfast and at bedtime, for a duration of 3 months.
  Interventions: Combination Product: Steroid nasal drops combined with olfactory training
- Placebo Nasal Drops Combined with Olfactory Training Group (Placebo Comparator): The placebo group will receive normal saline nasal drops, with all other procedures identical to those in the intervention group.
  Interventions: Combination Product: Placebo nasal drops combined with olfactory training

INTERVENTIONS:
Combination Product: Steroid nasal drops combined with olfactory training — The intervention consists of two components: steroid nasal drops and modified olfactory training.
  Arms: Hormone Nasal Drops Combined with Olfactory Training Group
Combination Product: Placebo nasal drops combined with olfactory training — The intervention consists of two components: normal saline nasal drops and modified olfactory training.
  Arms: Placebo Nasal Drops Combined with Olfactory Training Group

SUMMARY:
This study aims to evaluate the effectiveness of hormone nasal drops in the olfactory cleft combined with olfactory training for treating postinfectious olfactory dysfunction (PIOD). The main questions this clinical trial seeks to answer are:

Can the combination of hormone nasal drops and olfactory training improve smell function better than olfactory training alone in PIOD patients? How does this combined treatment work?

DETAILED DESCRIPTION:
Post-infectious olfactory dysfunction (PIOD) is a prevalent condition, particularly following viral upper respiratory infections such as COVID-19, and significantly impacts patients' quality of life. Current treatments primarily rely on olfactory training, but its effectiveness varies, with improvement rates ranging between 30% and 50%. Emerging evidence suggests that olfactory cleft obstruction and chronic inflammation play critical roles in PIOD pathogenesis, highlighting the potential benefits of targeted steroid therapy to address these underlying mechanisms.

In this study, the investigators planned to recruit 100 patients and divided them into two groups for combined therapy with steroid drops or placebo drops alongside olfactory training, and validate the effectiveness of the combined therapy based on the comparison of the outcomes of the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Prospective enrollment of otolaryngology clinic patients aged 18-65 years with olfactory dysfunction. Diagnosis of post-infectious olfactory dysfunction (PIOD) will be based on the PPOD 2023 criteria. Participants must demonstrate olfactory impairment via Sniffin' Sticks testing, with TDI scores (sum of Threshold, Discrimination, and Identification) meeting: (1) Hyposmia: 16 < TDI < 30.75; (2) Anosmia: TDI ≤ 15.
2. Willingness to participate and signed informed consent.

Exclusion Criteria:

1. Use of systemic corticosteroids within 4 weeks or intranasal steroids within 2 weeks prior to enrollment.
2. Severe nasal septum deviation, nasal tumors, acute upper respiratory infections, or uncontrolled allergic rhinitis.
3. History of functional endoscopic sinus surgery or other nasal procedures within 12 months.
4. Severe cardiovascular disease, hepatic/renal insufficiency, uncontrolled diabetes, or immune system disorders.
5. Current or planned pregnancy.
6. Investigator-determined inability to comply with study requirements (e.g., memory/behavioral disorders, depression, heavy alcohol use, prior non-compliance).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The Sniffin' Sticks test | Baseline, 1 week, 4 weeks, 8 weeks, and 12 weeks after the initiation of treatment.
  A clinically significant olfactory improvement as measured by Sniffin' Sticks threshold, discrimination, and identification(TDI)

SECONDARY OUTCOMES:
Questionnaire of Olfactory Disorders - Negative Statements (QOD-NS) | Baseline, 2 weeks, 4 weeks, 8 weeks, and 12 weeks after the initiation of treatment.
  The QOD-NS includes 17 negative statements, each graded from 0 (disagree) to 3 (agree) for a maximum score of 51. Higher QOD-NS scores reflect worse QoL.
Olfactory-Visual Analogue Scale (VAS) | Baseline, 2 weeks, 4 weeks, 8 weeks, and 12 weeks after the initiation of treatment.
  Subjects rate the impact of smell loss on their mood, ability to enjoy food, social interactions, safety, personal hygiene, sex life, ability to cook food, appetite and change in weight from 0 (no impact) to 10 (most impact) for a maximum score of 90. Higher olfactory-VAS scores reflect more severe impacts on daily life.
CT Evaluation of Olfactory Cleft Blockage | Baseline and 12 weeks after the initiation of treatment.
  The olfactory cleft was divided into anterior and posterior, divided by the anterior end of the superior turbinate. The anterior and posterior olfactory cleft opacifications were graded separately on a scale of 0-4 by the ratio of the opacified area to the whole area of the olfactory cleft, with 0 (no opacification),
  1 (25%), 2 (25%-50%), 3 (50%-75%), and 4 (>75%). The olfactory cleft CT score, calculated as the sum of the anterior and posterior olfactory cleft scores, ranged from 1 to 8 (Kim DW, Kim JY, Jeon SY. The status of the olfactory cleft may predict postoperative olfactory function in chronic rhinosinusitis with nasal polyposis. Am J Rhinol Allergy. 2011;25(2):e90-4.).
Inflammatory Marker Levels in Olfactory Mucosa | Baseline and 12 weeks after the initiation of treatment.
  Analysis of inflammatory cytokines （IL-4、IL-5、IL-13、IL-25、IL-33 and TSLP）via ELISA and single-cell sequencing from olfactory mucosal brush samples.
Plasma Cortisol Levels | Baseline and 12 weeks after the initiation of treatment.
  Measurement of systemic cortisol concentrations through venous blood sampling
Adverse Event | 2 weeks, and 4 weeks, 8 weeks, and 12 weeks after the initiation of treatment.
  Documentation of local (nasal irritation, epistaxis) and systemic steroid-related adverse events using standardized case report forms during all follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Dawei Wu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
We will decide whether to share the individual participant data after the study.